CLINICAL TRIAL: NCT00318955
Title: A Post-Marketing, Open-Label, Randomized, Comparative Study Comparing the Usefulness of Dexmedetomidine at the Time of Extubation and Post Extubation Period to Other Sedative Management in Post-Operative Patients
Brief Title: Post-Marketing Clinical Study to Assess Efficacy and Safety of Dexmedetomidine in Post-Operative Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Maruishi Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEX-401; NCT00248001 (obsolete NCT alias)
Record Dates: First submitted 2006-04-18; First posted 2006-04-27 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2015-06

CONDITIONS: Conscious Sedation
Keywords: Dexmedetomidine, Sedation, Extubation, Phase 4
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine group (Experimental)
  Interventions: Drug: Dexmedetomidine
- Propofol group (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: Dexmedetomidine group
Drug: Propofol
  Arms: Propofol group

SUMMARY:
The purpose of this study is to assess efficacy and safety of dexmedetomidine at the time of extubation and after extubation, in patients requiring postoperative sedation in the ICU.

DETAILED DESCRIPTION:
The study is to conduct as a phase IV post-marketing clinical study in accordance with the approval condition of dexmedetomidine hydrochloride in Japan. The study will compare the use of dexmedetomidine in patient management at the time of extubation with other sedative/ analgesic management, Comparison is made in the use of dexmedetomidine in patient management between a group in which management is performed with dexmedetomidine and a group in which standard management is performed with propofol in patients requiring postoperative sedation in the ICU The usefulness of dexmedetomidine during postextubation period is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally acceptable representative (if acceptable by Institutional Review Board/Ethics Committee) has signed and dated the Informed Consent after the study has been fully explained.
* Patient is male or female; at least 20 years of age.
* Patient who is in condition of American Society of Anesthesiology (ASA) I to III Class preoperatively
* Patient is orally intubated and anticipated to require sedation for mechanical ventilation for a minimum period of 4 hours following open-heart surgery, coronary artery bypass grafting (CABG), or major vascular surgery
* If patient is female with child bearing potential, she is to be non-pregnant, and not lactating

Exclusion Criteria:

* Patient with serious disturbance of the central nervous system (disturbance of consciousness).
* Patient has undergone or requires intracranial surgery during current hospitalization
* Patient requires muscle relaxant drugs after admission to the ICU (except when an endotracheal tube is reinserted).
* Patient requires epidural or intrathecal administration of analgesia/anesthesia after surgery and during their ICU stay.
* Patients for whom propofol or opioids are contraindicated.
* Patient has known or suspected allergies to any medication that might be administered during the course of the study.
* Patient is obese (body mass index >35)
* Patient was recently hospitalized for drug overdose
* Patient for whom alpha-2 antagonists or alpha-2 agonists are contraindicated
* Patient is currently or previously treated, within 30 days before the start of the study, with an alpha-2 antagonist or alpha-2 receptor agonist.
* Patient has participated in another clinical study within 30 days prior to admission to the ICU and patient is currently participating in another clinical study.
* Patient was diagnosed with severe symptoms and judged likely to die within 24 hours.
* Patient is considered unable to undergo all procedures required by the protocol.
* Patient with excessive bleeding that is likely require reoperation.
* Patient with an ejection fraction of < 30%.
* Patient, in the opinion of the investigator or subinvestigator in the post-marketing clinical study, that has symptoms or factors that may increase his/her risk as a result of the clinical study, or that may not provide sufficient study data.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2005-11; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who maintained a Richmond Agitation-Sedation score =0, -1, -2 | Continuously from 1 hour before extubation or end of propofol infusion before extubation, whichever is later, to 1 hour after extubation

SECONDARY OUTCOMES:
Variations in vital signs (blood pressure and heart rate) in patients | From 10 minutes before extubation to 10 minutes after extubation
Percentage of patients who required analgesia and received supplemental fentanyl before and after extubation | From 7 days prior to surgery to the start of surgery, and from the end of surgery to 48 hrs after the start of infusion
Percentage of patients with a total score of 3 on the Behavioral Pain Scale just before extubation | 10±2 minutes before extubation, 2±1 minutes after extubation
Percentage of patients who required supplemental sedation after extubation | After extubation to 24 hours after the start of study drug infusion.
Percentage of patients who require post-extubation analgesia and who received supplemental fentanyl after extubation | After extubation to 24 hours after the start of study drug infusion.
Amount of supplemental fentanyl required after extubation | After extubation to 24 hours after the start of study drug infusion.
Ratio of time with a Richmond Agitation-Sedation score ≥+1 | From 1 hour before extubation or the end of propofol infusion before extubation, whichever was later, to 1 hour after extubation
Distribution of Richmond Agitation-Sedation score most frequently recorded while intubated | From the start of study drug administration to 1 hour before the expected time of extubation.
Ease of patient management on the basis of a questionnaire to physicians and nurses | Conducted to the greatest possible extent, at ICU discharge or at 36 hours after the start of drug administration, whichever is earlier (in Part II only).
Assessment of interactions between dexmedetomidine and propofol or fentanyl | After propofol or fentanyl administration (Pre-dose and Post dose [5 and 10 minutes])
Patient self-evaluation of experiences during their stay in the ICU | Conducted to the greatest possible extent, at ICU discharge or at 36 hours after the start of drug administration, whichever is earlier (in Part II only).

CONTACTS AND LOCATIONS:
Overall Officials: Misa Kawai, Study Director — Hospira, now a wholly owned subsidiary of Pfizer
Locations (13):
- Japan (13):
  - Hirosaki University Hospital, Hirosaki-shi, Aomori
  - Kyushu University Hospital, Higashiku, Fukuoka
  - Kagoshima University Medical and Dental Hospital, Kagoshima, Kagoshima-ken
  - Kyoto University Hospital, Sakyoku, Kyoto
  - Nagasaki University Hospital of Medicine and Dentistry, Nagasaki, Nagasaki
  - Okayama University Hospital of Medicine and Dentistry, Okayama, Okayama-ken
  - Osaka City General Hospital, Miyakojima-ku, Osaka
  - Kinki University Hospital, Osaka-Sayama-Shi, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo

REFERENCES:
- [Background] Aitkenhead AR. Analgesia and sedation in intensive care. Br J Anaesth. 1989 Aug;63(2):196-206. doi: 10.1093/bja/63.2.196. No abstract available. PMID 2669909
- [Background] Minoru Kaneshiro. Analgesic and Sedatin during mechanical ventilation, ICU and CCU 14:14643-648,1990
- [Background] Syu Matsukawa, et.al.Sedation during ventilation control, ICU and CCU 14:603-608,1990
- [Background] Megumu Tagami et.al. Post-operative analgesic and sedation control,
- [Background] Greenblatt DJ, Divoll M, Abernethy DR, Ochs HR, Shader RI. Clinical pharmacokinetics of the newer benzodiazepines. Clin Pharmacokinet. 1983 May-Jun;8(3):233-52. doi: 10.2165/00003088-198308030-00003. PMID 6133664
- [Background] Hidekazu Yukioka, et.al. Current status of analgesic and sedation control in ICU. Japan ICU Treatment Association's Magazine 1:13-19, 1994
- [Background] Masayoshi Hyodo et.al. Anesthetic Science, 10th edition, Kinpodo, ppl 213-219
- [Background] Ikuto Yoshiya. Section 4; Pharmacology for Anesthesia, Introduction to Anesthesiology, 7th edition, Nagai Shoten,pp439-447, 1993
- [Background] Ikuto Yoshiya: Sedation and Analgesia for Intensive Care Patients. Anesthesia 21(2):2-6, 333-337, 2000
- [Background] Costas Katsanoulas. Concluding Remarks: Redefining Intensive Care Unit Sedation, International Congress and Symposium Series 221, 83-88
- [Background] Mantz,J., Singer,M. Importance of Patient Orientation and Rousability as Components of Intensive Care Unit Sedation, International Congress and Symposium Series 221, 23-29
- [Background] Hewitt PB. Subjective follow-up of patients from a surgical intensive therapy ward. Br Med J. 1970 Dec 12;4(5736):669-73. doi: 10.1136/bmj.4.5736.669. PMID 4098972